CLINICAL TRIAL: NCT02771990
Title: tDCS for Chronic Low Back Pain: A Study Examining the Effect of Transcranial Direct Current Stimulation on the Emotional Response to Chronic Low Back Pain
Brief Title: tDCS for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Benjamin Greenberg, Associate Director, CfNN, Providence VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-042
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Chronic Low Back Pain
Keywords: Back Pain
MeSH Terms: conditions — Back Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sham tDCS (Sham Comparator): 10 sessions sham transcranial direct current stimulation (tDCS)
  Interventions: Device: Sham transcranial direct current stimulation
- active tDCS (Experimental): 10 sessions active transcranial direct current stimulation (tDCS)
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: Sham transcranial direct current stimulation — sham stimulation
  Arms: sham tDCS
Device: transcranial direct current stimulation — 2 milliamp (mA) 20 minutes
  Arms: active tDCS

SUMMARY:
The goal of this study is to investigate the role of central neural pathways in mediating chronic pain. The aim of the study is to test the effect of stimulating brain regions that are part of a network underlying central pain processing using a non-invasive brain stimulation technique, transcranial Direct Current Stimulation (tDCS). Prior studies have used tDCS to target both sensory related cortical areas and those important for higher-order representations of pain. This study will target brain regions important for the behavioral response to the chronic sensation of pain. The hypothesis is that stimulation of these brain regions can modulate not only the affective component of pain, but ultimately also improve functioning and quality of life. This hypothesis will be tested by treating study participants eighteen and older with chronic low back pain (CLBP) of greater than six months using tDCS. To be part of this study, participants must meet all the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Low Back Pain ≥ 6 months duration in the lumbar region, present more than half the days of the month, and on average be at a moderate level of severity in the last month
* At least one trial of physician recommended medication (e.g. acetaminophen, NSAIDS, skeletal muscle relaxants)
* Pre-existing opioid and non-opioid pain medication must be non-existent or stable (medications have not changed for one month)
* Be able to understand, read and write English
* If female and of childbearing age, agree to use acceptable birth control during the study treatment period (oral contraceptives, history of tubal ligation, history of a hysterectomy, or a reliable barrier method)

Exclusion Criteria:

* Lifetime Diagnostic and Statistical Manual (DSM) IV diagnosis of bipolar disorder, schizophrenia, or other chronic psychotic condition
* Current DSM-IV diagnosis of substance dependence for alcohol, sedative/hypnotic drugs, stimulants, cocaine
* Current cancer, infection, or inflammatory arthritis
* Broken skin or other lesions in the area of the electrodes
* Uncontrolled medical problems, such as diabetes mellitus, hypertension, pulmonary or airway disease, heart failure, coronary artery disease, or any other condition that poses a risk for the subject during participation
* Presence of metal in the cranial cavity
* Holes in the skull made by trauma or surgery
* Pacemakers, medication pumps, and other implanted electronic hardware
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Burgess, MD, PhD, Principal Investigator — Providence VA Medical Center; Benjamin Greenberg, MD, PhD, Principal Investigator — Providence VA Medical Center

IPD SHARING:
Plan to Share IPD: No
Only de-identified data will be shared.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 30 participants that were consented, 9 participants were ineligible, withdrew, or were lost to contact before commencing tDCS.
Period: Overall Study
Arm/Group | Sham tDCS | Active tDCS
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham tDCS | Active tDCS | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (1.8) | 65.7 (8.8) | 63.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 9 | 9 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 7 | 14
  Black or African American | 1 | 0 | 1
  Hispanic or Latino | 0 | 1 | 1
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Other | 3 | 2 | 5
Years of Education [Mean (Standard Deviation); unit: years] | 14.7 (2.6) | 14.0 (2.6) | 14.4 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: West Haven-Yale Multidimensional Pain Inventory (WHY-MPI) General Activity Subscale Rating
Description: The WHY-MPI General Activity subscale contains 18 items summed to give a score ranging from 0 to 108 (higher scores indicate more activity [better]).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sham tDCS: 10 sessions sham transcranial direct current stimulation (tDCS)
  Sham transcranial direct current stimulation: sham
Arm/Group | Sham tDCS | Active tDCS
Number analyzed (Participants) | 11 | 10
score on a scale | 35.3 (17.7) | 48.4 (21.2)
Statistical Analysis 1: Comparison: Sham tDCS vs Active tDCS; Test type: Other — Pilot study; p = 0.002, Regression, Linear; z-score = 3.11

2. Primary Outcome: Pain Anxiety Symptom Scale (PASS-20) Rating
Description: The PASS-20 contains 20 items and scores could range from 0 to 100 (higher scores indicate greater pain anxiety).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham tDCS | Active tDCS
Number analyzed (Participants) | 11 | 10
score on a scale | 26.4 (22.0) | 26.3 (23.6)
Statistical Analysis 1: Comparison: Sham tDCS vs Active tDCS; Test type: Other — Pilot study; p = 0.67, Regression, Linear

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Sham tDCS: 10 sessions sham transcranial direct current stimulation (tDCS)
  Sham transcranial direct current stimulation: sham stimultion
Arm/Group | Sham tDCS | Active tDCS
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
small sample size (N = 21), participants were not stratified by premorbid anxiety levels, inability to guarantee optimal targeting of the left dorsal anterior cingulate cortex, inability to address laterality effects of pain perception

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT02771990/Prot_SAP_000.pdf